CLINICAL TRIAL: NCT01044888
Title: Heparin Resistance During Off-pump Coronary Artery Bypass Graft Surgery: Predictors and Clinical Implication
Brief Title: Heparin Resistance: Predictors and Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2007-0142
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Off Pump Coronary Artery Bypass Surgery
Keywords: Heparin responsiveness; Off-pump coronary artery bypass graft surgery; Risk factors; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Heparin — 150 U/kg heparin was administered intravenously at the beginning of graft anastomosis and accepted a perioperative ACT value of around 300 s. Ten minutes after the loading dose, the ACT was measured. An ACT of 300 s or greater was considered as adequate. Then follow up ACT measurement was determined after 30 min from the previous ACT measurement. If ACT fell below the target value of 300 s, an additional dose of heparin was administered. If ACT was between 250 and 299 s, additional 2000 U of heparin was administered and if ACT was between 200 and 249 s then additional 3000 U of heparin was injected. Ten minutes after additional heparin injection, ACT was remeasured.

SUMMARY:
The investigators evaluated clinical impact of reduced heparin responsiveness (HRreduced) on the incidence of perioperative myocardial infarction (MI) and restenosis at 6 months after off-pump coronary artery bypass graft surgery (OPCAB) and identified its predictors.

ELIGIBILITY:
Inclusion Criteria:

* enrolling all consecutive patients scheduled for elective isolated multivessel OPCAB between April 2007 and March 2008

Exclusion Criteria:

* presence of known preoperative coagulopathy, emergency operation or preoperative use of an intra-aortic balloon pump.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
incidences of postoperative MI and major morbidity | immediate postoperative period

SECONDARY OUTCOMES:
incidences of cardiac morbidities | 6 months following surgery
restenosis of graft vessels | 6 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hee Chun, MD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance hospital, Seoul, Seodaemungu, South Korea